CLINICAL TRIAL: NCT02674659
Title: The Effect of Resistance Training on Proprotein Subtilisin Convertase Kexin 9 (PCSK-9) Level in Patients After Coronary Bypass Surgery
Brief Title: The Effect of Resistance Training on Proprotein Subtilisin Convertase Kexin 9 Level After Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Bambang Dwiputra, MD, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RUHK-2016
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
Keywords: resistance training, PCSK9, coronary artery bypass grafting
MeSH Terms: conditions — Coronary Artery Disease; Hypercholesterolemia, Autosomal Dominant, 3 | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Patients after coronary bypass surgery who undergo conventional cardiac rehabilitation program (aerobic training only)
  Interventions: Behavioral: aerobic training
- Intervention group (Experimental): Patients after coronary bypass surgery who undergo conventional cardiac rehabilitation program plus resistance training (aerobic and resistance training as well)
  Interventions: Behavioral: resistance training; Behavioral: aerobic training

INTERVENTIONS:
Behavioral: resistance training — resistance training consists of lower and upper extremities exercises. We focus on biceps and hamstring to be trained. One session was held for around 30 minutes.
  Arms: Intervention group
Behavioral: aerobic training — aerobic exercise consists of warming up session, treadmill exercise (around 20-30 minutes), and wrap-up session (for all session about 1 hour)

SUMMARY:
This research add resistance training to patients who undergo cardiac rehabilitation program after coronary bypass surgery, comparing the level of PCSK9 level on that group to another group who receives conventional rehabilitation program (only aerobic exercise)

DETAILED DESCRIPTION:
The PCSK9 level measured before and after cardiac rehabilitation program (around 3-4 weeks), and compared between two groups. ELISA method will be used to measure plasma PCSK9 level.

Resistance training will be given by professional trainer in gymnasium of National Cardiovascular Center Harapan Kita supervised by cardiologists, following rules from American College of Sports Medicine guideline regarding to exercise after cardiac event.

ELIGIBILITY:
Inclusion Criteria:

* post elective coronary artery bypass surgery
* > 18 years old
* sign informed consent

Exclusion Criteria:

* contraindications of resistance training (unstable angina, uncontrolled blood pressure (systolic > 160 mmHg diastolic > 100 mmHg), acute heart failure, pulmonary diseases, arrhythmia malignant)
* musculoskeletal pain, visual analog scale >3
* post congenital heart disease surgery
* post elective coronary artery bypass surgery with malfunction valves (operated or not)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Dwiputra, MD, Principal Investigator — National Cardiovascular Center Harapan Kita

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor RS, Brown A, Ebrahim S, Jolliffe J, Noorani H, Rees K, Skidmore B, Stone JA, Thompson DR, Oldridge N. Exercise-based rehabilitation for patients with coronary heart disease: systematic review and meta-analysis of randomized controlled trials. Am J Med. 2004 May 15;116(10):682-92. doi: 10.1016/j.amjmed.2004.01.009. PMID 15121495
- [Background] Cornelissen VA, Fagard RH, Coeckelberghs E, Vanhees L. Impact of resistance training on blood pressure and other cardiovascular risk factors: a meta-analysis of randomized, controlled trials. Hypertension. 2011 Nov;58(5):950-8. doi: 10.1161/HYPERTENSIONAHA.111.177071. Epub 2011 Sep 6. PMID 21896934
- [Result] Ghroubi S, Elleuch W, Abid L, Abdenadher M, Kammoun S, Elleuch MH. Effects of a low-intensity dynamic-resistance training protocol using an isokinetic dynamometer on muscular strength and aerobic capacity after coronary artery bypass grafting. Ann Phys Rehabil Med. 2013 Mar;56(2):85-101. doi: 10.1016/j.rehab.2012.10.006. Epub 2012 Dec 7. PMID 23414745
- [Result] Busch JC, Lillou D, Wittig G, Bartsch P, Willemsen D, Oldridge N, Bjarnason-Wehrens B. Resistance and balance training improves functional capacity in very old participants attending cardiac rehabilitation after coronary bypass surgery. J Am Geriatr Soc. 2012 Dec;60(12):2270-6. doi: 10.1111/jgs.12030. Epub 2012 Nov 23. PMID 23176104
- [Result] Kamani CH, Gencer B, Montecucco F, Courvoisier D, Vuilleumier N, Meyer P, Mach F. Stairs instead of elevators at the workplace decreases PCSK9 levels in a healthy population. Eur J Clin Invest. 2015 Oct;45(10):1017-24. doi: 10.1111/eci.12480. Epub 2015 Aug 26. PMID 26081791
- [Result] Urban D, Poss J, Bohm M, Laufs U. Targeting the proprotein convertase subtilisin/kexin type 9 for the treatment of dyslipidemia and atherosclerosis. J Am Coll Cardiol. 2013 Oct 15;62(16):1401-8. doi: 10.1016/j.jacc.2013.07.056. Epub 2013 Aug 21. PMID 23973703
- [Result] Kim HS, Wu Y, Lin SJ, Deerochanawong C, Zambahari R, Zhao L, Zhang Q, Yan P. Current status of cholesterol goal attainment after statin therapy among patients with hypercholesterolemia in Asian countries and region: the Return on Expenditure Achieved for Lipid Therapy in Asia (REALITY-Asia) study. Curr Med Res Opin. 2008 Jul;24(7):1951-63. doi: 10.1185/03007990802138731. Epub 2008 Jun 10. PMID 18547466
- [Result] Sullivan D, Olsson AG, Scott R, Kim JB, Xue A, Gebski V, Wasserman SM, Stein EA. Effect of a monoclonal antibody to PCSK9 on low-density lipoprotein cholesterol levels in statin-intolerant patients: the GAUSS randomized trial. JAMA. 2012 Dec 19;308(23):2497-506. doi: 10.1001/jama.2012.25790. PMID 23128163
- [Result] Cohen JC, Boerwinkle E, Mosley TH Jr, Hobbs HH. Sequence variations in PCSK9, low LDL, and protection against coronary heart disease. N Engl J Med. 2006 Mar 23;354(12):1264-72. doi: 10.1056/NEJMoa054013. PMID 16554528
- [Result] Lagace TA, Curtis DE, Garuti R, McNutt MC, Park SW, Prather HB, Anderson NN, Ho YK, Hammer RE, Horton JD. Secreted PCSK9 decreases the number of LDL receptors in hepatocytes and in livers of parabiotic mice. J Clin Invest. 2006 Nov;116(11):2995-3005. doi: 10.1172/JCI29383. PMID 17080197
- [Result] Zhang DW, Lagace TA, Garuti R, Zhao Z, McDonald M, Horton JD, Cohen JC, Hobbs HH. Binding of proprotein convertase subtilisin/kexin type 9 to epidermal growth factor-like repeat A of low density lipoprotein receptor decreases receptor recycling and increases degradation. J Biol Chem. 2007 Jun 22;282(25):18602-18612. doi: 10.1074/jbc.M702027200. Epub 2007 Apr 23. PMID 17452316
- [Result] Wen S, Jadhav KS, Williamson DL, Rideout TC. Treadmill Exercise Training Modulates Hepatic Cholesterol Metabolism and Circulating PCSK9 Concentration in High-Fat-Fed Mice. J Lipids. 2013;2013:908048. doi: 10.1155/2013/908048. Epub 2013 Jun 19. PMID 23862065
- [Result] European Association of Cardiovascular Prevention and Rehabilitation Committee for Science Guidelines; EACPR; Corra U, Piepoli MF, Carre F, Heuschmann P, Hoffmann U, Verschuren M, Halcox J; Document Reviewers; Giannuzzi P, Saner H, Wood D, Piepoli MF, Corra U, Benzer W, Bjarnason-Wehrens B, Dendale P, Gaita D, McGee H, Mendes M, Niebauer J, Zwisler AD, Schmid JP. Secondary prevention through cardiac rehabilitation: physical activity counselling and exercise training: key components of the position paper from the Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur Heart J. 2010 Aug;31(16):1967-74. doi: 10.1093/eurheartj/ehq236. Epub 2010 Jul 19. PMID 20643803
- [Result] Fiorina C, Vizzardi E, Lorusso R, Maggio M, De Cicco G, Nodari S, Faggiano P, Dei Cas L. The 6-min walking test early after cardiac surgery. Reference values and the effects of rehabilitation programme. Eur J Cardiothorac Surg. 2007 Nov;32(5):724-9. doi: 10.1016/j.ejcts.2007.08.013. Epub 2007 Sep 18. PMID 17881241
- [Result] Wang J, Yu W, Zhao D, Liu N, Yu Y. In-Hospital and Long-Term Mortality in 35,173 Chinese Patients Undergoing Coronary Artery Bypass Grafting in Beijing: Impact of Sex, Age, Myocardial Infarction, and Cardiopulmonary Bypass. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):26-31. doi: 10.1053/j.jvca.2016.08.004. Epub 2016 Aug 4. PMID 27771273
- [Result] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Result] Pieri M, Belletti A, Monaco F, Pisano A, Musu M, Dalessandro V, Monti G, Finco G, Zangrillo A, Landoni G. Outcome of cardiac surgery in patients with low preoperative ejection fraction. BMC Anesthesiol. 2016 Oct 18;16(1):97. doi: 10.1186/s12871-016-0271-5. PMID 27760527
- [Result] Abifadel M, Varret M, Rabes JP, Allard D, Ouguerram K, Devillers M, Cruaud C, Benjannet S, Wickham L, Erlich D, Derre A, Villeger L, Farnier M, Beucler I, Bruckert E, Chambaz J, Chanu B, Lecerf JM, Luc G, Moulin P, Weissenbach J, Prat A, Krempf M, Junien C, Seidah NG, Boileau C. Mutations in PCSK9 cause autosomal dominant hypercholesterolemia. Nat Genet. 2003 Jun;34(2):154-6. doi: 10.1038/ng1161. PMID 12730697
- [Result] Careskey HE, Davis RA, Alborn WE, Troutt JS, Cao G, Konrad RJ. Atorvastatin increases human serum levels of proprotein convertase subtilisin/kexin type 9. J Lipid Res. 2008 Feb;49(2):394-8. doi: 10.1194/jlr.M700437-JLR200. Epub 2007 Nov 21. PMID 18033751
- [Result] Boyer M, Levesque V, Poirier P, Marette A, Mathieu P, Despres JP, Larose E, Arsenault BJ. Impact of a 1-year lifestyle modification program on plasma lipoprotein and PCSK9 concentrations in patients with coronary artery disease. J Clin Lipidol. 2016 Nov-Dec;10(6):1353-1361. doi: 10.1016/j.jacl.2016.08.014. Epub 2016 Sep 2. PMID 27919352
- [Result] Baass A, Dubuc G, Tremblay M, Delvin EE, O'Loughlin J, Levy E, Davignon J, Lambert M. Plasma PCSK9 is associated with age, sex, and multiple metabolic markers in a population-based sample of children and adolescents. Clin Chem. 2009 Sep;55(9):1637-45. doi: 10.1373/clinchem.2009.126987. Epub 2009 Jul 23. PMID 19628659
- [Result] Chen YW, Hubal MJ, Hoffman EP, Thompson PD, Clarkson PM. Molecular responses of human muscle to eccentric exercise. J Appl Physiol (1985). 2003 Dec;95(6):2485-94. doi: 10.1152/japplphysiol.01161.2002. Epub 2003 Aug 22. PMID 12937035
- [Result] Brooks N, Layne JE, Gordon PL, Roubenoff R, Nelson ME, Castaneda-Sceppa C. Strength training improves muscle quality and insulin sensitivity in Hispanic older adults with type 2 diabetes. Int J Med Sci. 2006 Dec 18;4(1):19-27. doi: 10.7150/ijms.4.19. PMID 17211497
- [Result] Arsenault BJ, Pelletier-Beaumont E, Almeras N, Tremblay A, Poirier P, Bergeron J, Despres JP. PCSK9 levels in abdominally obese men: association with cardiometabolic risk profile and effects of a one-year lifestyle modification program. Atherosclerosis. 2014 Oct;236(2):321-6. doi: 10.1016/j.atherosclerosis.2014.07.010. Epub 2014 Jul 26. PMID 25128757
- [Result] Shaibi GQ, Cruz ML, Ball GD, Weigensberg MJ, Salem GJ, Crespo NC, Goran MI. Effects of resistance training on insulin sensitivity in overweight Latino adolescent males. Med Sci Sports Exerc. 2006 Jul;38(7):1208-15. doi: 10.1249/01.mss.0000227304.88406.0f. PMID 16826016
- [Result] Kelley GA, Kelley KS. Progressive resistance exercise and resting blood pressure : A meta-analysis of randomized controlled trials. Hypertension. 2000 Mar;35(3):838-43. doi: 10.1161/01.hyp.35.3.838. PMID 10720604
- [Derived] Dwiputra B, Santoso A, Purwowiyoto BS, Radi B, Ambari AM. The effect of resistance training on PCSK9 levels in patients undergoing cardiac rehabilitation after coronary artery bypass grafting: a randomized study. BMC Cardiovasc Disord. 2023 Nov 9;23(1):549. doi: 10.1186/s12872-023-03571-7. PMID 37946122
- See also: website of hospital where the study protocol will be held — http://www.pjnhk.go.id/
- See also: website of educational institution inside the hospital — http://www.ui.ac.id

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We initiate this project from February 10th, 2016 until September 23rd, 2016. All the subjects (post coronary artery bypass graft operation) were collected from the National Cardiovascular Center Harapan Kita.
Pre-assignment Details: There is no specific run-in period for every patient enrolled in this study. If they meet the inclusion criteria, they will be randomly assigned to the intervention or control group.
Groups:
- Intervention Group: Patients after coronary bypass surgery who undergo conventional cardiac rehabilitation program plus resistance training (aerobic and resistance training as well)
  resistance training: resistance training consists of lower and upper extremities exercises. We focus on biceps and hamstring to be trained. One session will be held for around 15 minutes.
  aerobic training: aerobic exercise consists of warming up session, treadmill exercise (around 20-30 minutes), and wrap-up session (for all session about 1 hour)
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 43 | 44
Completed | 39 | 40
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Customized [Mean (Standard Deviation); unit: years old]
  Age | 57.2 (8.4) | 56.3 (8.1) | 56.8 (8.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex : Sex | 43 | 44 | 87
  Sex : Male | 38 | 39 | 77
  Sex : Female | 5 | 5 | 10
Height [Mean (Standard Deviation); unit: cm] | 164.5 (6.8) | 162.9 (6.4) | 163.7 (6.6)
weight [Mean (Standard Deviation); unit: kg] | 68.2 (10.6) | 65.9 (10.9) | 67.1 (10.8)
waist circumference [Mean (Standard Deviation); unit: cm] | 97.5 (10.5) | 95.1 (10.8) | 96.3 (10.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (2.9) | 24.6 (3.1) | 24.9 (3)
Cardiovascular risk factor [Count of Participants; unit: Participants]
  Hypertension | 32 | 31 | 63
  Diabetes Mellitus | 20 | 21 | 41
  Dyslipidemia | 21 | 21 | 42
  Smoking | 32 | 33 | 65
  Family history | 6 | 8 | 14
Ejection Fraction [Mean (Standard Deviation); unit: %] | 52.1 (15.2) | 50.2 (15.4) | 51.1 (15.3)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 121.1 (14.8) | 125.3 (17.9) | 123.2 (16.4)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.5 (9.8) | 76.8 (9.9) | 75.7 (9.9)
Statin therapy [Count of Participants; unit: Participants]
  Simvastatin | 32 | 33 | 65
  Simvastatin 10 mg | 4 | 3 | 7
  Simvastatin 20 mg | 28 | 30 | 58
  Atorvastatin | 11 | 11 | 22
Length of stay [Mean (Standard Deviation); unit: days] | 9.1 (4.0) | 9.1 (3.9) | 9.1 (4.0)
CPB duration [Mean (Standard Deviation); unit: minutes] — Population: CABG patients on pump (using CPB machine)
  minutes
    number analyzed (Participants) | 38 | 40 | 78
    (all) | 81.5 (26.4) | 81.2 (21.3) | 81.4 (23.9)
Aortic cross clamp duration [Mean (Standard Deviation); unit: minutes] — Population: CABG patients on pump (using CPB machine)
  minutes
    number analyzed (Participants) | 38 | 40 | 78
    (all) | 48.9 (24.1) | 47.6 (16.9) | 48.3 (20.5)
Cardiac Rehabilitation Program Type [Count of Participants; unit: Participants]
  Frequency 3 times/week | 18 | 20 | 38
  Frequency 5 times/week | 25 | 24 | 49
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 116.5 (41.5) | 116.6 (37.6) | 116.6 (39.6)
Lipid profile [Mean (Standard Deviation); unit: mg/dL]
  Total Cholesterol | 161.1 (32.4) | 160.4 (36.5) | 160.8 (34.5)
  High Density Lipoprotein | 32.9 (8.5) | 34.5 (8.0) | 33.7 (8.3)
  Low Density Lipoprotein | 96.7 (30.1) | 96.3 (30.2) | 96.5 (30.2)
  Trigliseride | 172.2 (63.2) | 171.8 (58.7) | 172 (70)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: mg/dL] | 24.6 (16.5) | 28.8 (16.6) | 26.7 (16.6)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: mg/dL] | 44.3 (23.3) | 49.2 (24.2) | 46.8 (23.8)
Uric acid [Mean (Standard Deviation); unit: mg/dL] | 7.1 (1.1) | 7.1 (1.6) | 7.1 (1.4)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.07 (0.3) | 1.03 (0.2) | 1.05 (0.3)
PCSK-9 [Mean (Standard Deviation); unit: ng/ml] | 382.4 (127.3) | 407.04 (112.3) | 394.7 (119.8)

OUTCOME MEASURES:

1. Primary Outcome: PCSK-9 Level
Description: this outcome measurement will be achieved by taking patient's blood sample after cardiac rehabilitation program. The method that we use to check PCSK-9 level is ELISA method
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Population: Patients who completed the cardiac rehabilitation program
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 39 | 40
ng/ml | 377.5 (118.9) | 322.53 (107.5)

2. Secondary Outcome: Low Density Lipoprotein
Description: this outcome measurement will be achieved by taking patient's blood sample after cardiac rehabilitation program
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 43 | 44
mg/dL | 106.3 (26.6) | 96.2 (24.9)

3. Secondary Outcome: Body Mass Index
Description: Body Mass Index is calculated by calculating the measured body weight divided by the height square in measure. We take BMI data after cardiac rehabilitation program in every participant.
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 43 | 44
kg/m^2 | 25.3 (2.9) | 24.7 (3.0)

4. Secondary Outcome: High-Density Lipoprotein
Description: this outcome measurement will be achieved by taking patient's blood sample after cardiac rehabilitation program
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 43 | 44
mg/dL | 36.1 (7.0) | 37.4 (7.9)

5. Secondary Outcome: Total Cholesterol
Description: this outcome measurement will be achieved by taking patient's blood sample after cardiac rehabilitation program
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 43 | 44
mg/dL | 162.2 (32.6) | 162.1 (35.5)

6. Secondary Outcome: Triglyceride
Description: This outcome measurement will be achieved by taking the patient's blood sample after cardiac rehabilitation program
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 43 | 44
mg/dL | 145.7 (50.2) | 139.4 (50.7)

7. Secondary Outcome: Fasting Blood Glucose
Description: Blood glucose concentration was taken after 10-12-hour fasting. This outcome measurement will be achieved by taking the patient's blood sample after cardiac rehabilitation program
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 43 | 44
mg/dL | 107.7 (24.6) | 102.4 (22.9)

8. Secondary Outcome: Systolic Blood Pressure
Description: this outcome measurement will be achieved by taking the patient's blood pressure after cardiac rehabilitation program
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 43 | 44
mmHg | 117.3 (11.4) | 118.8 (12.5)

9. Secondary Outcome: Diastolic Blood Pressure
Description: this outcome measurement will be achieved by taking the patient's blood pressure after cardiac rehabilitation program
Time Frame: 3-4 weeks (after completion of 12 sessions of cardiac rehabilitation program)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 43 | 44
mmHg | 73.8 (6.3) | 74.8 (10.3)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/44
Other Adverse Events (participants affected / at risk) | 2/43 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=43) | Intervention Group (N=44)
Acute heart failure (Cardiac disorders) | 1 (1) | 1 (1) — acute decompensated heart failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=43) | Intervention Group (N=44)
wound infection (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — postoperative wound infection

LIMITATIONS AND CAVEATS:
This study only investigated selected population of patients (post CABG patients) and cannot explain further the mechanism of reduced PCSK9 level by doing resistance training

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No